CLINICAL TRIAL: NCT01839890
Title: Study to Evaluate the Efficacy and Safety of Paclitaxel Eluting Balloon in St Elevation Myocardial Infarction After Bare Metal Stent Insertion
Brief Title: Paclitaxel Eluting Balloon in St Elevation Myocardial Infarction
Acronym: PEBSI-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Francisco Javier Goicolea (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor-Investigator, Francisco Javier Goicolea, Dr. Fco. Javier Goicolea, Fundación Médica para la Investigación y Desarrollo en el Area Cardiovascular
Organization: Fundación Médica para la Investigación y Desarrollo en el Area Cardiovascular (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PEBSI-01
Record Dates: First submitted 2013-03-26; First posted 2013-04-25 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2014-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Paclitaxel; stent; Acute infarction; Systolic time elevation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bare metal Stent plus Paclitaxel Balloon (Experimental): Conventional bare metal Stent plus Paclitaxel Eluting Balloon(Pantera Lux)®
  Interventions: Device: Bare metal Stent plus Paclitaxel Balloon
- Bare metal Stent (Active Comparator): Conventional Bare Stent
  Interventions: Device: Bare metal Stent

INTERVENTIONS:
Device: Bare metal Stent plus Paclitaxel Balloon — After the permeabilization of the clinical event responsible artery with conventional therapy (including the insertion of a conventional metal stent and once by the interventional cardiologist gives good final result), patients will be randomized in a 1:1 ratio
  Other Names: Balloon PANTERA LUX (R)
  Arms: Bare metal Stent plus Paclitaxel Balloon
Device: Bare metal Stent — After the permeabilization of the clinical event responsible artery with conventional therapy a conventional metal stent will be inserted. Once by the interventional cardiologist gives good final result), patients will be randomized in a 1:1 ratio
  Other Names: PROKINETIC ENERGY (R)
  Arms: Bare metal Stent

SUMMARY:
Study objective is the evaluation of safety and efficacy at 9 months of combination treatment of bare metal Stent plus Paclitaxel Eluting Balloon vs bare metal stent (conventional treatment) in patients with acute myocardial infarction with systolic time elevation of less than 12 hours of evolution.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open study

After the permeabilization of the clinical event responsible artery and the insertion of a bare metal stent, patients will be randomized in a 1:1 ratio to one of the following treatment groups:

Group 1: post-dilatation with a paclitaxel eluting balloon (Pantera Lux ®) Group 2: no post-dilatation Patients (or their legal representative) must sign the consent before randomization.

After surgery, patients will be treated with dual antiplatelet therapy (aspirin plus clopidogrel) for at least one month to group 2 patients; and at least 3 months in those who are also treated with the paclitaxel eluting balloon (group 1). Aspirin is prescribed indefinitely according to the usual practice in these patients.

Patients will be monitored 30 days after surgery, at 6 and 12 months, and the ninth month (in which patient will receive an angiographic control).

The primary efficacy endpoint is late lumen loss (PLT) comparing it value during surgery and control angiography at 9 months

This study will involve patients over 18 years olds with systolic time elevation myocardial infarction, or new left bundle branch block or posterior AMI (ECG) that occur within 12 hours of onset of symptoms to treatment by primary angioplasty.

They include a total of 220 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 18 years.
* Acute myocardial infarction (AMI) within 12 hours of evolution (from the onset of symptoms) systolic time elevation of at least 1 mm (recorded in two or more contiguous leads), new left bundle branch block, or true posterior infarction.
* Patients candidates for primary angioplasty as medical criteria
* Written informed consent according to International Conference on Harmonization / Guide Clinical Practice and local legislation, obtained before any study procedure.
* Diameter vascular coronary artery to treat between 2 mm and 4 mm.
* Patients with 90-100% stenosis.

Exclusion Criteria:

* Patients who refuse to participate in the study
* Cardiogenic shock (defined as systolic blood pressure less than 80 mm Hg for more than 30 minutes or need for vasopressors or intra-aortic balloon counterpulsation)
* Concomitant diseases associated with a life expectancy of less than one year
* Angiographic variables:

  * Trunk unprotected
  * Branching (side branch greater than 2.5 mm)
  * Sinus tachycardia segment elevation myocardial infarction thrombosis secondary to stent
  * If more than one stent to treat a single segment (overlapping stents).
  * Patient candidate for surgical revascularization within 30 days
  * Stenosis of greater than 30 mm in length (corresponding with the ball longer available)
  * Reference vessel diameter less than 2.5 mm and greater than 4 mm (larger ball)
  * More severe stenosis in the same artery in which is expected to be addressed in the next 9 months
* Women at childbearing age, where there is the possibility of pregnancy during the first year of follow-up, or nursing.
* Any clinical condition, which in the opinion of the investigator, is considered clinically significant as to participate in the study.
* Subjects who are participating in any study drug or medical.
* Individuals who show inability to follow instructions or help during the course of the study.
* Bleeding diathesis or other disorders such as gastrointestinal ulceration or cerebral circulatory disorders, restricting the use of treatments platelet aggregation inhibitors and anticoagulants.
* Patients with an ejection fraction <30% (if known).
* Allergy or hypersensitivity to paclitaxel intolerance, or compounds structurally related to the Butyryl tri-n-hexyl citrate (BTHC) matrix of administration.
* Severe allergy to contrast media.
* Coronary artery spasm in the absence of significant stenosis.
* Cases in which is indicated bypass surgery within 30 days after infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Late Luminal Loss | 1 year
  Loss measured in millimeters of late luminal space in vessels

SECONDARY OUTCOMES:
Efficacy | 1 year
  Efficacy: angiography restenosis, minimal luminal diameter, ischemia directed target vessel revascularization (TVR), MACE (death, infarction, TVR)
Safety | 1 year
  Safety: MACE/ month, at 6 months and 12 months (death, re-infarction, acute cardiovascular disease, hemorrhagy and/or stent thrombosis).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Goicolea, PhD, Study Director — Hospital Universitario Puerta de Hierro. Majadahonda. Madrid
Locations (19):
- Spain (19):
  - Complexo Hospitalario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Albacete, Albacete, Albacete
  - H. Regional Universitario Infanta Cristina, Badajoz, Badajoz
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario Valle de Hebrón, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres, Cáceres
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Regional Universitario Carlos Haya, Málaga, Málaga
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Galdakao-Usanso, Galdakao, Vizcaya

REFERENCES:
- [Derived] Garcia-Touchard A, Sabate M, Gonzalo N, Peral V, Vaquerizo B, Ruiz-Salmeron R, Garcia Del Blanco B, Jimenez-Mazuecos J, Molina E, Martinez-Romero P, Hernandez-Garcia JM, Ruiz-Quevedo V, Urbano C, Fernandez-Portales J, Rumoroso JR, Casanova-Sandoval J, Pinar E, Lopez-Pais J, Oteo JF, Alfonso F. Very long-term efficacy and safety of paclitaxel-eluting balloon after a bare-metal stent for the treatment of ST-elevation myocardial infarction: 8-year results of a randomized clinical trial (PEBSI study). Cardiovasc Diagn Ther. 2023 Oct 31;13(5):792-804. doi: 10.21037/cdt-22-623. Epub 2023 Oct 17. PMID 37941845